CLINICAL TRIAL: NCT03873077
Title: Effect of Local Infiltration Analgesia on Postoperative Pain Following Anterior Cruciate Ligament Reconstruction
Brief Title: Effect of LIA on Postoperative Pain Following ACL Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Dr. Alain Kalmar, MD, PhD, Staff Anesthesist, Algemeen Ziekenhuis Maria Middelares
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MMS.2019.001
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Anterior Cruciate Ligament Rupture; Pain, Postoperative
Keywords: local infiltration analgesia; postoperative analgesia
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Group A receives standard treatment (intravenous analgesia). Group B received intravenous analgesia and a LIA.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intravenous analgesia (No Intervention): Patient receives intravenous analgesia: paracetamol 30 mg/kg, diclofenac 75 mg, clonidine 1 µg/kg and morfine 0,05 mg/kg
- intravenous analgesia + LIA (Other): Patient receives intravenous analgesia and a local infiltration analgesia in the knee
  Interventions: Procedure: local infiltration analgesia

INTERVENTIONS:
Procedure: local infiltration analgesia — 10 mL ropivacaine 7.5 mg/mL and 10 mL lidocaine 10 mg/mL
  Arms: intravenous analgesia + LIA

SUMMARY:
An anterior cruciate ligament (ACL) rupture is one of the most common sport injuries, which typically develops after a sudden knee torsion. Arthroscopic repair of the ACL is often required as a complete ACL tear can cause instability of the knee joint.

During arthroscopic reconstruction the lower leg is reattached to the upper leg using part of the hamstring tendon (mm. gracilis and mm. semitendinosus). Optimal postoperative analgesia is necessary to allow a quick recovery. Intravenous analgesia during surgery is often associated with a number of side effects such as nausea, vomiting and muscle weakness and does not anesthetize the donor site of the hamstring tendon graft. Local infiltration of ropivacaine and lidocaine in the knee joint and at the donor site can be a valuable asset to control the postoperative pain.

This study evaluates the effect of local infiltration analgesia (LIA) on the postoperative pain in the first month after an ACL reconstruction. Half of participants will only receive intravenous analgesia during surgery, the other half will receive intravenous analgesia and a LIA.

DETAILED DESCRIPTION:
2 x 20 patients which are planned for arthroscopic ACL reconstruction are randomised: standard-group and LIA-group.

All patients receive standardised multimodal intravenous analgesia. After standardised induction of anesthesia, patient positioning and administration of basic analgetics (paracetamol, diclofenac, clonidine and morfine), patients in the LIA-group receive a local infiltration in the knee of 10 mL ropivacaine and 10 mL lidocaine.

Visual Analogue Scores are assessed 15 minutes after awakening from surgery and on Day 1, 2, 3, 7, 14, 21 and 28 after surgery. Postoperative analgesic consumption are registered in the first month after the surgery. The quality of recovery after anesthesia is assessed on Day 1 by the postoperative quality of recovery score (QoR-15).

ELIGIBILITY:
Inclusion Criteria:

* elective arthroscopic anterior cruciate ligament reconstruction
* adult

Exclusion Criteria:

* unwilling or unable to grant written informed consent
* revisions
* contra-indication for ropivacaine

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale for pain | From moment of surgery until one month after surgery
  Pain intensity using the VAS (where 0 = no pain and 100 = pain as bad as can be) 15 minutes after awakening and on Day 1, 2, 3, 7, 14, 21 and 28 after surgery.

SECONDARY OUTCOMES:
Postoperative analgesia consumption | From moment of surgery until one month after surgery
  Dosing and frequency of analgesia consumption
General patient comfort | From moment of surgery until one day after surgery
  Quality of recovery score (QoR-15) on the first day after surgery
Incidence of nausea and vomiting | From moment of surgery until hospital discharge (one day after surgery)
  Incidence of postoperative nausea and vomiting
PONV treatment | From moment of surgery until hospital discharge (one day after surgery)
  Number of pharmacological treatments for postoperative nausea and vomiting (PONV)

CONTACTS AND LOCATIONS:
Overall Officials: Alain F Kalmar, Principal Investigator — Maria Middelares Hospital
Locations (1):
- General Hospital Maria Middelares, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Background] Lefevre N, Klouche S, de Pamphilis O, Herman S, Gerometta A, Bohu Y. Peri-articular local infiltration analgesia versus femoral nerve block for postoperative pain control following anterior cruciate ligament reconstruction: Prospective, comparative, non-inferiority study. Orthop Traumatol Surg Res. 2016 Nov;102(7):873-877. doi: 10.1016/j.otsr.2016.07.011. Epub 2016 Oct 4. PMID 27720193
- [Background] Kerr DR, Kohan L. Local infiltration analgesia: a technique for the control of acute postoperative pain following knee and hip surgery: a case study of 325 patients. Acta Orthop. 2008 Apr;79(2):174-83. doi: 10.1080/17453670710014950. PMID 18484242
- [Background] Kristensen PK, Pfeiffer-Jensen M, Storm JO, Thillemann TM. Local infiltration analgesia is comparable to femoral nerve block after anterior cruciate ligament reconstruction with hamstring tendon graft: a randomised controlled trial. Knee Surg Sports Traumatol Arthrosc. 2014 Feb;22(2):317-23. doi: 10.1007/s00167-013-2399-x. Epub 2013 Jan 23. PMID 23338666